CLINICAL TRIAL: NCT02803151
Title: A Prospective Phase II Clinical Trial of Stereotactic Ablative Radiotherapy for Metastatic Lymphadenopathy
Brief Title: A Clinical Trial of Stereotactic Ablative Radiotherapy for Metastatic Lymphadenopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201601023RINA
Record Dates: First submitted 2016-06-06; First posted 2016-06-16 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Metastasis of Malignant Neoplasm to Lymph Node
Keywords: Stereotactic ablative radiotherapy; Lymph node metastasis; T cell immunity; cell-free DNA
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic ablative radiotherapy (Experimental): Image-guided stereotactic ablative radiotherapy
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — SABR with 36 to 45 Gy in six fractions to the defined target volume with met organ-at-risk constraint criteria using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc). Treatment should be given once per day, 2-3 fractions per week with no more than 2 consecutive daily fractions, over 2 to 2.5 weeks.
  Other Names: Stereotactic body radiotherapy; Hypofractionated image-guided radiotherapy

SUMMARY:
Lymph node metastasis is one of the most common sites to develop disease recurrence or progression after initial local treatment for primary solid malignancies or systemic treatment for advanced metastases. No specific treatment modality has been established as the standard therapy. Systemic therapy is usually considered since lymphadenopathy is considered as a sign of disease dissemination though aggressive local treatment, including surgical lymphoadenectomy or radical radiotherapy might result in long-term survival in selected patients. The concept of stereotactic ablative radiotherapy (SABR), a high dose of radiation targeted to a pathological entity and delivered in a few fractions, has proven so successful at treating both benign and malignant lesions that it changed the paradigm for radiation therapy. The radiobiology of SABR has been shown to be very favorable for tumor control. Clinical experiences suggested that SABR might offer excellent in-field tumor control with low toxicity profile in selected patients, although the majority of reports are retrospective and include small patients series with heterogeneous tumor sites and dose-fractionation schedules.

At present, there is lack of validated prognostic factors to identify the patients who might benefit most from ablative local therapy for metastatic lymph node(s). The mechanism of effect of SABR on the cancer lesions is not yet clear. Apart from its direct effect on clonogenic cancer cells, an immune-mediated process was also hypothesized. Therefore, the present study is aimed to provide a better understanding about utilization of SABR for metastatic lymph node(s). The associated translational researches will also advance our knowledge in the immune system reactions to SABR.

DETAILED DESCRIPTION:
This is a single institutional, single-arm, phase II trial to assess the local control rate of oligo-metastatic or oligo-progressive lymph node treated by stereotactic ablative radiotherapy at 1 year.

Patients with pathologically proven non-hematopoietic malignancy patients with radiographic evidence of evaluable regional recurrent, oligo-metastatic or oligo-progressive lymph nodes are eligible for enrolment.

Stereotactic Ablative Radiotherapy:

The lymph node planning target volume (PTV) will receive the prescribed dose according to the assigned treatment group. The dose is prescribed such as 90-95% of PTV is covered by the prescription dose. If the critical structures exceed the defined dose limitation, a dose reduction method is applied as protocol defined. Dose inhomogeneity can exist within the clinical target volume (CTV).

Treatment will be delivered in six fractions to the target volume and given once per day, 2-3 fractions per week with no more than 2 daily consecutive fractions, over 2 to 2.5 weeks.

Target Radiation Dose: SABR with 45 Gy in six fractions to the defined target volume with met organ-at-risk constraint criteria using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).

Radiation Dose Reduction:

Reduced Dose 10%: SABR with 40.05 Gy in six fractions to the defined target volume with met organ-at-risk constraint criteria

Reduced Dose 20%: SABR with 36 Gy in six fractions to the defined target volume with met organ-at-risk constraint criteria

ELIGIBILITY:
Inclusion criteria

1. Patients with a histologic diagnosis of non-hematopoietic malignancy
2. Radiographic evidence of measurable enlarged metastatic lymph node(s) with short-axis ≥ 1 cm
3. Patients do not have prior radiotherapy to the index node(s)
4. Age ≥ 20 years
5. Karnofsky performance status (KPS) ≥ 60%.
6. Life expectancy of ≥ 4 month
7. Patients must have adequate renal function with serum creatinine ≤ 2.0 mg/dL measured within 90 days prior to registration
8. Women of childbearing potential and male participants must practice adequate contraception
9. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion criteria

1. Prior radiotherapy to the index metastatic lymph node(s)
2. Sum of the greatest dimensions of index lymph note(s) exceed 6 cm
3. Inability to achieve the minimal required radiation dose (36Gy)
4. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration
   3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   7. Uncontrolled psychiatric disorder
5. Will receive any other investigational agent or chemotherapy and/or target therapies during treatment
6. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Local control (Response Evaluation Criteria In Solid Tumors version 1.1) | 12 months
  Number of participant with local progression of index metastatic lymph receiving stereotactic ablative radiotherapy, assessed on CT scan according to Response Evaluation Criteria In Solid Tumors version 1.1

SECONDARY OUTCOMES:
Patient reported outcome (Quality of Life questionnaire) | at 1, 3 months after radiotherapy, and every 3 month thereafter until unequivocal progression, hospice care, or death, assessed up to 12 months
  EORTC Quality of Life-Core 30 questionnaire module
Acute toxicity (Common Toxicity Criteria for Adverse Events version 4) | From date of radiotherapy until 90 days after radiotherapy starts
  Common Toxicity Criteria for Adverse Events version 4
Late toxicity (Common Toxicity Criteria for Adverse Events version 4) | From 90 days after radiotherapy starts until the date of death from any cause, up to 60 months
  Common Toxicity Criteria for Adverse Events version 4
Metastatic nodal progression | From date of enrolment until the date of first documented metastatic nodal progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participant with nodal progression on CT scan
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
  Number of participant alive

OTHER OUTCOMES:
Changes of peripheral blood lymphocyte subpopulations | at baseline, 2 weeks, 1, 2, 3, 6, and 12 months after radiotherapy
  T-cell subpopulation (CD3/4/8/19/16+56)

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Tapei, Taiwan

IPD SHARING:
Plan to Share IPD: No